CLINICAL TRIAL: NCT00522314
Title: Airway Clearance in Bronchiectasis: is Non-Invasive Ventilation a Useful Adjunct in Moderate to Severe Disease?A Pilot Study.
Brief Title: Airway Clearance in Bronchiectasis: is Non-Invasive Ventilation a Useful Adjunct in Moderate to Severe Disease?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1233R020
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Bronchiectasis
Keywords: Non-invasive ventilation; Airway clearance; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): NIV & ACBT
  Interventions: Device: NIV and ACBT
- 2 (Placebo Comparator): Active cycle of breathing techniques
  Interventions: Other: Active Cycle of Breathing Techniques

INTERVENTIONS:
Device: NIV and ACBT
  Arms: 1
Other: Active Cycle of Breathing Techniques
  Arms: 2

SUMMARY:
This clinical trial is investigating the efficacy of Non Invasive Ventilation (NIV) as a method of airway clearance in patients with an acute exacerbation and moderate to severe bronchiectasis disease. Current treatment focuses on the use of Active Cycle of Breathing Techniques (ACBT) but this modality alone may not be sufficient when patients have more severe disease and an acute infection. The use of NIV may result in better patient care and more appropriate physiotherapy treatment in the more unwell population.The aim of this study is to compare the efficacy of two physiotherapy airways clearance interventions in bronchiectasis.

DETAILED DESCRIPTION:
Twenty patients with moderate to severe bronchiectasis admitted to hospital with an acute exacerbation were recruited (October 2004 to April 2006) and allocated to one of two groups that received twice daily airway clearance treatment for a course of IVAB. Group 1 {ACBT} and group 2 {NIV and ACBT}. A number of measurements were recorded on the first and final day of treatment as well as daily to provide important comparative information on physiological changes, ease of use, and clinical efficacy.

Outcomes measured on day 1 and final day of IVAB were: LifeshirtTM which recorded tidal volume; respiratory rate; airway flow; thoracoabdominal coordination; oxygen saturation and heart rate during treatment; respiratory muscle strength (PImax and PEmax); spirometry; arterial blood gases (ABGs); breathlessness scores; patients perception of tiredness, benefit and ease of treatment; auscultation; number of coughs per treatment; duration of treatment; sputum production, wet and dry weight; sputum rheology.

The Lifeshirt is a novel technique (respiratory induction plethysmography)which provides data on a wide range of dynamic lung function values (lung volumes; flow volume curves; relative excursion of rib cage and abdomen; SpO2) during airway clearance intervention to help understanding of the possible mechanisms of action of different airway clearance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe bronchiectasis (FEV1 < 60%),
* Indicators of difficulty expectorating sputum, and
* An acute exacerbation requiring intravenous antibiotics (IVAB)

Exclusion Criteria:

* Unable to tolerate positive pressure
* Presence of pneumothorax

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | Before; mid-way; on completion of intravenous antibiotics

SECONDARY OUTCOMES:
Sputum weight | During airway clearance; half hour after airway clearance; 24 hour sputum clearance
Breathlessness | Before and after each airway clearance session
respiratory mechanics (Vivometrics Lifeshirt) | On first and last airway clearance session

CONTACTS AND LOCATIONS:
Overall Officials: Prof Elborn, MD, Principal Investigator — Belfast City Hospital and Queens University Belfast
Locations (1):
- Belfast City Hospital, Belfast, Northern Ireland, United Kingdom